CLINICAL TRIAL: NCT00832611
Title: A Study of the Effect of the ROX Percutaneous Arteriovenous Fistula System (ROX AC1) on Exercise Capacity and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study of the Effect of the ROX AC1 on Exercise Capacity and Quality of Life in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ROX Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROX IX
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung Disease; Chronic Airflow Obstruction; Chronic Bronchitis; Chronic Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Bronchitis, Chronic | interventions — Arteriovenous Shunt, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Group A Anastomotic Coupler (Experimental): Device: ROX Anastomotic Coupler System (ACS). The ACS will be used to create an arteriovenous fistula in the iliac region (between the iliac artery and vein).
  Interventions: Device: Arteriovenous Fistula (ROX AC1)

INTERVENTIONS:
Device: Arteriovenous Fistula (ROX AC1) — The percutaneous creation of an arteriovenous fistula.

SUMMARY:
To demonstrate the efficacy of ROX AC1 (with respect to exercise capacity and quality of life) in patients with COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic disease that leads to irreversible changes in the lung structure, but also to systemic changes in the body that can influence the severity of the disease. The irreversible changes to the lungs can be seen in limitations in the pulmonary function. The purpose of this clinical investigation is to evaluate the performance and efficacy of the ROX AC1 on exercise capacity and respiratory quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced Chronic Obstructive Pulmonary Disease (COPD) must be made on the basis of current findings, medical history and physical examination.

Exclusion Criteria:

* Subject not qualifying because of physical or psychological condition that may put them at risk of participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Improvement in exercise capacity. | 12 weeks post-procedure

SECONDARY OUTCOMES:
Improvement in quality of life. | 12 weeks post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Claus Vogelmeier, MD, Principal Investigator — Universitätsklinikum Gieβen und Marburg, Standort Marburg
Locations (1):
- Universitätsklinikum Gieβen und Marburg, Standort Marburg, Marburg, Germany

REFERENCES:
- [Background] Cooper CB, Celli B. Venous admixture in COPD: pathophysiology and therapeutic approaches. COPD. 2008 Dec;5(6):376-81. doi: 10.1080/15412550802522783. PMID 19353352
- [Derived] Faul J, Schoors D, Brouwers S, Scott B, Jerrentrup A, Galvin J, Luitjens S, Dolan E. Creation of an iliac arteriovenous shunt lowers blood pressure in chronic obstructive pulmonary disease patients with hypertension. J Vasc Surg. 2014 Apr;59(4):1078-83. doi: 10.1016/j.jvs.2013.10.069. Epub 2014 Jan 28. PMID 24484754